CLINICAL TRIAL: NCT06637306
Title: Pilot Trial of the IL-4 Receptor Antagonist Dupilumab Plus Pembrolizumab, Paclitaxel, and Carboplatin in Locally Advanced Triple Negative Breast Cancer
Brief Title: Neoadjuvant Dupilumab, Pembrolizumab, Paclitaxel, and Carboplatin in Locally Advanced Triple Negative Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rima Patel (Other)
Responsible Party: Sponsor-Investigator, Rima Patel, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRMC-24-125
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Triple Negative Breast Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: Dupilumab; Pembrolizumab; IL-4 Receptor Antagonist; Breast Cancer; Triple Negative; Locally Advanced
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — dupilumab; pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Open Label, Single Arm Trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with locally advanced TNBC (Experimental): Patients with advanced triple negative breast cancer (TNBC).
  Interventions: Drug: Dupilumab; Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Dupilumab — Dupilumab 600mg subcutaneous initial loading dose, 300mg for subsequent doses; administered every 3 weeks for 4 cycles. Immunotherapy drug FDA approved to treat patients with eczema, asthma, chronic rhinosinusitis with nasal polyps, and eosinophilic esophagitis. Investigational/not yet FDA approved to treat patients with breast cancer.
  Other Names: DUPIXENT
Drug: Pembrolizumab — Pembrolizumab 200mg intravenous every 3 weeks for 4 cycles and one 400mg intravenous dose one week following completion of chemotherapy. Cancer immunotherapy drug FDA approved for the treatment of high-risk, early-stage, triple-negative breast cancer (TNBC).
  Other Names: KEYTRUDA
Drug: Paclitaxel — Paclitaxel 80mg/m2 intravenous weekly for 12 weeks. Chemotherapy FDA-approved for the treatment of patients with breast cancer.
  Other Names: TAXOL
Drug: Carboplatin — Carboplatin AUC 1.5 intravenous weekly for 12 weeks. Chemotherapy FDA-approved for the treatment of patients with breast cancer.

SUMMARY:
Pilot trial of the IL-4 receptor antagonist dupilumab plus pembrolizumab, paclitaxel, and carboplatin in locally advanced triple negative breast cancer (TNBC).

Primary Objective: To assess the safety of neoadjuvant dupilumab and pembrolizumab plus weekly paclitaxel and carboplatin as measured by the proportion of severe immune-related adverse events (irAEs) in patients with locally advanced TNBC.

Secondary Objectives: To determine the rates of pathologic complete response with the addition of dupilumab to NAC and pembrolizumab; to determine the rate of residual cancer burden 0-1; to estimate the recurrence-free survival and overall survival; to assess the toxicity of the combination of dupilumab, pembrolizumab, and paclitaxel-carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed diagnosis of triple negative breast cancer, as defined by the most recent ASCO/CAP guidelines.
* Patients must have previously untreated, localized TNBC with either tumor size ≥ 2 centimeters (T2-4N0) or lymph node involvement with at least a 1cm tumor (T1c-T4N1-3).
* Patients must have previously untreated disease with no prior definitive breast surgery, radiation therapy, or systemic chemotherapy with therapeutic intent for this breast cancer.
* Patients must be eligible to receive chemotherapy agents in the study including paclitaxel and carboplatin.
* Patients must be willing and able to provide blood samples at the time points indicated in the study calendar.
* Patients must be willing and able to have core needle biopsies of tumor prior to initiation of treatment. Should patients undergo pre-treatment or on-treatment biopsy procedure and inadequate number of biopsies are obtained, they may proceed with initiation/continuation of treatment at the discretion of the investigator and treating physician.
* Age ≥ 18 years.
* ECOG performance status 0-1.
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or any treatment with therapeutic intent for the breast cancer.
* Patients may not be receiving any other investigational agents.
* Patients who have any distant metastases and considered to have Stage IV disease.
* Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Patients with active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, paclitaxel, dupilumab or pembrolizumab used in study. Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps).
* HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <350 CD4+ T cells/microliter in the peripheral blood.
* Known active Hepatitis B (e.g., HBV detected by PCR or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
* Known, untreated helminth infections. Patients with prior history of a helminth infection who were fully treated are permitted.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine within 30 days of planned start of study medication.
* History of irAE in response to prior immunotherapy that has not improved to a Grade 0 or 1; this does not include chronic conditions such as endocrinopathies which can be treated with hormone replacement therapy.
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis attributed to prior use of cancer immunotherapy that required immune-suppressive doses of glucocorticoids to assist with management. History of radiation pneumonitis treated with glucocorticoids.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe immune-related adverse events (irSAE) | Within 4 months of therapy
  Incidence of severe immune-related adverse events within 4 months of therapy.
  Immune related Severe Adverse Events (irSAE) are defined as:
  * Any Grade 4 immune-related AE with the exception of hypothyroidism
  * Any Grade 3 immune-related AE requiring permanent discontinuation of dupilumab and pembrolizumab
  * Any new Grade 3 or Grade 4 non-hematologic laboratory abnormality, if
    * medical intervention is required, or
    * the abnormality leads to hospitalization, or
    * the abnormality persists for > 72 hours
  * Any non-hematologic AE which is considered severe or life-threatening and requires discontinuation of dupilumab and pembrolizumab
  * Any ≥ Grade 2 immune-mediated uveitis
  * Any immune-related AE resulting in persistent or significant disability/incapacity (substantial disruption of one's ability to conduct normal life functions) for a period of 30 days or greater
  * Grade 5 or life-threatening toxicity

SECONDARY OUTCOMES:
Proportion of patients with pathologic complete response (pCR) with 95 percent Wilson Score interval | During procedure, after 13 weeks of neoadjuvant therapy
  Pathologic complete response (pCR) is defined as the lack of invasive cancer in the breast and axilla at time of surgical resection after neoadjuvant therapy. The research team will calculate the proportion of patients with pathologic complete response with 95 percent Wilson Score interval without continuity correction.
Proportion of patients with residual cancer burden (RCB) categories 0 and 1 with 95 percent Wilson Score | After completion of neoadjuvant therapy (13 weeks)
  Residual cancer burden (RCB) categories 0-1 comprise of patients who have achieved pCR (RCB 0) and have minimal tumor burden (RCB 1) after neoadjuvant therapy. The research team will calculate the proportion of patients with residual cancer burden categories 0 and 1 with 95 percent Wilson Score interval without continuity correction.
Proportion of patients who did not experience an invasive breast cancer recurrence (Recurrence-Free Survival (RFS)) | During procedure, after 13 weeks of neoadjuvant therapy
  Recurrence-free survival (RFS) is measured as the proportion of patients who did not experience an invasive breast cancer recurrence in the ipsilateral breast or regional nodes, distant organ sites, or death from any cause for the specified time period. It is defined as time from start of treatment to occurrence of an invasive breast cancer recurrence in the ipsilateral breast or regional nodes, distant organ sites, or death from any cause.
  The research team will summarize using Kaplan-Meier method with 95 percent pointwise confidence intervals using complimentary log-log scale. Median RFS with 95 percent confidence interval will be calculated using Brookmeyer and Crowley method. Hazard ratios with 95 percent confidence interval will be estimated using Proportional Hazards Cox regression model.
Overall Survival (OS) | After completion of neoadjuvant therapy (13 weeks)
  Overall survival (OS) is defined as the time from the start of treatment until documented death from any cause. The research team will summarize using Kaplan-Meier method with 95 percent pointwise confidence intervals using complimentary log-log scale. Median RFS with 95 percent confidence interval will be calculated using Brookmeyer and Crowley method. Hazard ratios with 95 percent confidence interval will be estimated using the Cox Proportional Hazards regression model.
Number of immune-related adverse events grades 3-5 | Within 3 months and 6 months of treatment
  Toxicity will be measured by the number immune-related adverse events grades 3-5 and incidence of severe TEAE (Grade 3-5 or serious AEs) according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, as well as based on rates of dose interruptions and drug discontinuations due to adverse events.
Number of adverse events measured using CTCAE Version 5.0 | Within 3 months and 6 months of treatment
  Number of adverse events will be reported according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of all-grade immune-related adverse events | Within 3 months and 6 months of treatment
  Incidence of all-grade immune-related adverse events and severe TEAEs with the combination therapy within 3 months at the last study visit and within 6 months with chart review.
Type of adverse events | Within 3 months and 6 months of treatment
  The type of severe adverse events will be collected.
Number of dose interruptions | Within 3 months and 6 months of treatment
  The research team will assess the number of dose interruptions due to AEs with 95 percent Wilson Score interval without continuity correction.
Number of drug discontinuations | Within 3 months and 6 months of treatment
  The research team will assess the number of drug discontinuations due to AEs with 95 percent Wilson Score interval without continuity correction.

CONTACTS AND LOCATIONS:
Overall Officials: Rima Patel, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Joseph Sparano, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Contact the Sponsor-Investigator via email: Rima.Patel2@mssm.edu